CLINICAL TRIAL: NCT02896712
Title: Developing Adaptive Interventions for Cocaine Cessation and Relapse Prevention ("Adaptive Trial")
Brief Title: Developing Adaptive Interventions for Cocaine Cessation and Relapse Prevention
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Joy Schmitz, Professor and CNRA Director, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSC-MS-15-0595
Record Dates: First submitted 2016-09-06; First posted 2016-09-12 (Estimated); Results first posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Cocaine-Related Disorders
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Acceptance and Commitment Therapy; Starch; Modafinil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- ACT plus CM (Active Comparator): Acceptance and Commitment Therapy along with Contingency Management for cocaine use will be administered to help decrease experiential avoidance while increasing acceptance and willingness to experience unpleasant thoughts, feelings, and physical symptoms.
  Interventions: Behavioral: Acceptance and Commitment Therapy (ACT); Behavioral: Contingency Management (CM)
- ACT plus CM, with Placebo (Active Comparator): Acceptance and Commitment Therapy along with Contingency Management for cocaine use will be administered and augmented with a placebo capsule during Phase 2 (weeks 5-12).
  Interventions: Behavioral: Acceptance and Commitment Therapy (ACT); Behavioral: Contingency Management (CM); Drug: Placebo
- ACT plus CM, with Modafinil (Experimental): Acceptance and Commitment Therapy along with Contingency Management for cocaine use will be administered and augmented with a Modafinil (300mg) capsule during Phase 2 (weeks 5-12).
  Interventions: Behavioral: Acceptance and Commitment Therapy (ACT); Behavioral: Contingency Management (CM); Drug: Modafinil
- DC plus CM (Active Comparator): Drug Counseling and Contingency Management for cocaine use will be administered to help educate patients about important concepts in addiction recovery.
  Interventions: Behavioral: Drug Counseling (DC); Behavioral: Contingency Management (CM)
- DC plus CM, with Placebo (Active Comparator): Drug Counseling and Contingency Management for cocaine use will be administered and augmented with a placebo capsule during Phase 2 (weeks 5-12).
  Interventions: Behavioral: Drug Counseling (DC); Behavioral: Contingency Management (CM); Drug: Placebo
- DC plus CM, with Modafinil (Experimental): Drug Counseling and Contingency Management for cocaine use will be administered and augmented with a Modafinil (300mg) capsule during Phase 2 (weeks 5-12).
  Interventions: Behavioral: Drug Counseling (DC); Behavioral: Contingency Management (CM); Drug: Modafinil

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy (ACT) — ACT will assist cocaine patients to notice internal cravings and triggers, abandon attempts to manage these triggers via active avoidance, suppression or other control-based strategies, and to make commitments to engage in behaviors consistent with chosen values or goals. ACT encourages clients to experience thoughts and feelings from an observer perspective, and helps clients not to believe distressing thoughts and feelings as if those thoughts and feelings are literally true and in need of action. ACT treatment will be based on the ACT therapy manual developed and tested previously.
  Other Names: ACT
  Arms: ACT plus CM; ACT plus CM, with Modafinil; ACT plus CM, with Placebo
Behavioral: Drug Counseling (DC) — The investigators will use the manual-guided individual DC modeled after the NIDA Collaborative Cocaine Treatment Study and used as the active control therapy in previous studies. DC approximates clinical practice as it is considered the most common type of evidence-based treatment in the community for patients actively using cocaine.
  Other Names: DC
  Arms: DC plus CM; DC plus CM, with Modafinil; DC plus CM, with Placebo
Behavioral: Contingency Management (CM) — The investigators will use the same high-magnitude CM schedule shown previously to be feasible and effective in facilitating initial cocaine abstinence. Subjects will earn vouchers for cocaine-negative urine samples collected at scheduled clinic visits each week. Under an escalating reinforcement schedule, voucher values will begin at $15 and increase by $10 for each consecutive negative urine. Bonus vouchers of $10 will be given for three consecutive negative urines. Provision of a cocaine-positive urine or failure to provide a scheduled sample will result in no vouchers earned and will reset the schedule to the initial value of $15.
  Other Names: CM
Drug: Placebo — The placebo capsule will be filled with corn starch and riboflavin.
  Other Names: Corn Starch
  Arms: ACT plus CM, with Placebo; DC plus CM, with Placebo
Drug: Modafinil — Modafinil capsules will start at 200 mg (day 1) and increase to the fixed dose of 300 mg (day 2) and will also contain riboflavin.
  Other Names: Provigil
  Arms: ACT plus CM, with Modafinil; DC plus CM, with Modafinil

SUMMARY:
First, the investigators will determine whether Acceptance and Commitment Therapy in combination with Contingency Management increases initial treatment response rates.

Second, for patients who do not respond to initial treatment, the investigators will examine whether dopamine-targeted pharmacotherapy is an effective augmentation strategy.

Third, for patients who respond to initial treatment, the investigators will assess the relative benefit of continued treatment with Acceptance and Commitment Therapy in combination with Contingency Management, as compared to Drug Counseling in combination with Contingency Management, to prevent relapse.

DETAILED DESCRIPTION:
Drug addiction is a chronic, devastating, but treatable disorder, for which there exists a growing armamentarium of evidence-based interventions, including pharmacotherapies and psychotherapies. A core principle of drug addiction treatment, however, states that no single treatment is appropriate for everyone; rather, treatments need to be adjusted based on patient characteristics and response in order to be maximally effective. Ideally, clinicians would identify a sequence of interventions that works best across different stages of addiction treatment, from abstinence initiation to relapse prevention. Adaptive treatment interventions have been used successfully to inform this sequential clinical decision-making process. For cocaine use disorders (CUD), the most potent intervention currently available for initiating abstinence is behavior therapy using contingency management (CM) procedures. Intensive CM has been shown to produce initial cocaine abstinence rates of 40%, unmatched by all other forms of behavioral or pharmacological treatment, making it a prototypical first-line therapy for CUD. Importantly, achievement of initial abstinence predicts future abstinence. For the clinician, these research findings translate into a straightforward question: Can the investigators drive CM response rates even higher with targeted adjunctive interventions?

The proposed sequential, multiple assignment, randomized trial (SMART) will provide the data needed to answer this question. First, the investigators will determine whether Acceptance and Commitment Therapy (ACT) in combination with CM increases initial treatment response rates. The investigators hypothesize that four weeks of treatment with ACT+CM will produce higher abstinence rates than initial treatment combining standard Drug Counseling with CM (DC+CM). The hypothesized synergism of ACT+CM on primary treatment mechanisms of experiential avoidance and reward sensitivity, respectively, will be examined. Second, for patients who do not respond to initial treatment, the investigators will examine whether dopamine-targeted pharmacotherapy is an effective augmentation strategy. Specifically, the investigators hypothesize that continued ACT+CM treatment with modafinil augmentation will be most effective in promoting abstinence relative to treatment combinations involving continued DC and/or placebo. Third, for patients who respond to initial treatment, the investigators will assess the relative benefit of continued treatment with ACT+CM, as compared to DC+CM, to prevent relapse. ACT emphasizes goal-directed actions based on values that are intrinsically motivating, and is thereby expected to be a more effective intervention for extending the duration of abstinence following initial treatment with intensive CM.

ELIGIBILITY:
Inclusion Criteria:

1. be between 18 and 60 years of age
2. meet DSM-5 criteria for current cocaine use disorder of at least moderate severity (≥ 4 symptoms)
3. have at least 1 positive urine BE specimen (≥ 150 ng/mL) during intake
4. be in acceptable health on the basis of interview, medical history and physical exam
5. agree to use an acceptable method of birth control during study participation and for one month after discontinuation of the study medication. Non-hormonal methods of contraception are recommended, including barrier contraceptives (e.g., diaphragm, cervical cap, male condom) or intrauterine device (IUD). Steroid contraceptives if used with non-hormonal methods are acceptable.
6. be able to understand the consent form and provide written informed consent
7. be able to provide the names of at least 2 persons who can generally locate their whereabouts.

Exclusion Criteria:

1. current DSM-5 diagnosis for substance use disorder (of at least moderate severity) other than cocaine, marijuana, or nicotine
2. have a DSM-5 axis I psychiatric disorder or neurological disease or disorder requiring ongoing treatment and/or making study participation unsafe (e.g., psychosis, dementia).
3. significant current suicidal or homicidal ideation
4. medical conditions contraindicating modafinil pharmacotherapy (e.g., major cardiovascular disease, severe liver disease based on Child-Pugh score of B or C, serious kidney problems)
5. taking medications that could adversely interact with modafinil (e.g., propranolol, phenytoin, warfarin, diazepam)
6. having conditions of probation or parole requiring reports of drug use to officers of the court
7. impending incarceration
8. pregnant or nursing for female patients
9. inability to read, write, or speak English

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 118 (Actual)
Dates: Start 2016-11-18; Primary Completion 2021-09-13 (Actual); Study Completion 2021-09-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UTHealth Center for Neurobehavioral Research on Addiction, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Dios C, Webber HE, Wardle MC, Yoon JH, Patriquin MA, Vincent JN, Schmitz JM, Lane SD. Anti-saccade error rates are associated with somatic depressive symptoms in cocaine use disorder. J Psychopharmacol. 2025 Dec 26:2698811251399579. doi: 10.1177/02698811251399579. Online ahead of print. PMID 41451557
- [Derived] Nunez C, Yoon JH, de Dios C, Dang V, Lane SD, Vincent JN, Schmitz JM, Wardle MC. Undervaluing nondrug rewards or overvaluing cocaine? Cocaine demand relates to cocaine use severity more strongly than anhedonia in individuals with cocaine use disorder. Exp Clin Psychopharmacol. 2025 Feb;33(1):91-99. doi: 10.1037/pha0000744. Epub 2024 Aug 29. PMID 39207396
- [Derived] Webber HE, Yoon JH, de Dios C, Suchting R, Dang V, Versace F, Green CE, Wardle MC, Lane SD, Schmitz JM. Assessing cocaine motivational value: Comparison of brain reactivity bias toward cocaine cues and cocaine demand. Exp Clin Psychopharmacol. 2023 Aug;31(4):861-867. doi: 10.1037/pha0000622. Epub 2022 Dec 8. PMID 36480395
- [Derived] Lathan EC, Hong JH, Heads AM, Borgogna NC, Schmitz JM. Prevalence and Correlates of Sex Selling and Sex Purchasing among Adults Seeking Treatment for Cocaine Use Disorder. Subst Use Misuse. 2021;56(14):2229-2241. doi: 10.1080/10826084.2021.1981391. Epub 2021 Sep 24. PMID 34559026
- [Derived] Webber HE, de Dios C, Wardle MC, Suchting R, Green CE, Schmitz JM, Lane SD, Versace F. Electrophysiological responses to emotional and cocaine cues reveal individual neuroaffective profiles in cocaine users. Exp Clin Psychopharmacol. 2022 Oct;30(5):514-524. doi: 10.1037/pha0000450. Epub 2021 Feb 25. PMID 33630644
- [Derived] Yoon JH, Suchting R, McKay SA, San Miguel GG, Vujanovic AA, Stotts AL, Lane SD, Vincent JN, Weaver MF, Lin A, Schmitz JM. Baseline cocaine demand predicts contingency management treatment outcomes for cocaine-use disorder. Psychol Addict Behav. 2020 Feb;34(1):164-174. doi: 10.1037/adb0000475. Epub 2019 Jun 24. PMID 31233323

RESULTS

PARTICIPANT FLOW:
Groups:
- Acceptance and Commitment Therapy (ACT) Plus Contingency Management (CM) Only: This arm included participants who responded to ACT plus CM in phase 1, as well as participants who did not proceed to receive modafinil or placebo in phase 2.
  In phase 1 (weeks 1-4), ACT plus CM for cocaine use will be administered to help decrease experiential avoidance while increasing acceptance and willingness to experience unpleasant thoughts, feelings, and physical symptoms.
  In phase 2 (weeks 5-12), ACT plus CM for cocaine use will continue to be administered.
- ACT Plus CM, With Placebo: This arm included participants who did not respond to ACT plus CM in phase 1 and who proceeded to receive placebo in phase 2.
  In phase 1 (weeks 1-4), ACT plus CM for cocaine use will be administered to help decrease experiential avoidance while increasing acceptance and willingness to experience unpleasant thoughts, feelings, and physical symptoms.
  In phase 2 (weeks 5-12), ACT plus CM for cocaine use will continue to be administered and participants will also receive placebo.
- ACT Plus CM, With Modafinil: This arm included participants who did not respond to ACT plus CM in phase 2 and who proceeded to receive modafinil in phase 2.
  In phase 1 (weeks 1-4), ACT plus CM for cocaine use will be administered to help decrease experiential avoidance while increasing acceptance and willingness to experience unpleasant thoughts, feelings, and physical symptoms.
  In phase 2 (weeks 5-12), ACT plus CM for cocaine use will continue to be administered and participants will also receive modafinil.
- Drug Counseling (DC) Plus Contingency Management (CM) Only: This arm included participants who responded to DC plus CM in phase 1, as well as participants who did not proceed to receive modafinil or placebo in phase 2.
  In phase 1 (weeks 1-4), DC plus CM for cocaine use will be administered to help educate patients about important concepts in addiction recovery.
  In phase 2 (weeks 5-12), DC plus CM for cocaine use will continue to be administered.
- DC Plus CM, With Placebo: This arm included participants who did not respond to DC plus CM in phase 1 and who proceeded to receive placebo in phase 2.
  In phase 1 (weeks 1-4), DC plus CM for cocaine use will be administered to help educate patients about important concepts in addiction recovery.
  In phase 2 (weeks 5-12), DC plus CM for cocaine use will continue to be administered and participants will also receive placebo.
- DC Plus CM, With Modafinil: This arm included participants who did not respond to DC plus CM in phase 1 and who proceeded to receive modafinil in phase 2.
  In phase 1 (weeks 1-4), DC plus CM for cocaine use will be administered to help educate patients about important concepts in addiction recovery.
  In phase 2 (weeks 5-12), DC plus CM for cocaine use will continue to be administered and participants will also receive modafinil.
Period: Phase 1
Arm/Group | Acceptance and Commitment Therapy (ACT) Plus Contingency Management (CM) Only | ACT Plus CM, With Placebo | ACT Plus CM, With Modafinil | Drug Counseling (DC) Plus Contingency Management (CM) Only | DC Plus CM, With Placebo | DC Plus CM, With Modafinil
Started | 18 | 17 | 19 | 21 | 23 | 20
Completed | 14 | 17 | 19 | 10 | 23 | 20
Not Completed | 4 | 0 | 0 | 11 | 0 | 0
Period: Phase 2
Arm/Group | Acceptance and Commitment Therapy (ACT) Plus Contingency Management (CM) Only | ACT Plus CM, With Placebo | ACT Plus CM, With Modafinil | Drug Counseling (DC) Plus Contingency Management (CM) Only | DC Plus CM, With Placebo | DC Plus CM, With Modafinil
Started | 14 | 17 | 19 | 10 | 23 | 20
Completed | 8 | 11 | 10 | 9 | 13 | 13
Not Completed | 6 | 6 | 9 | 1 | 10 | 7

BASELINE CHARACTERISTICS:
Groups:
- Phase 1: ACT Plus CM: Acceptance and Commitment Therapy along with Contingency Management for cocaine use will be administered to help decrease experiential avoidance while increasing acceptance and willingness to experience unpleasant thoughts, feelings, and physical symptoms.
- Phase 1: DC Plus CM: Drug Counseling and Contingency Management for cocaine use will be administered to help educate patients about important concepts in addiction recovery.
- Total: Total of all reporting groups
Arm/Group | Phase 1: ACT Plus CM | Phase 1: DC Plus CM | Total
Number analyzed (Participants) | 54 | 64 | 118
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.48 (8.74) | 51.58 (6.58) | 49.7 (7.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 42 | 52 | 94
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 6 | 12
  Not Hispanic or Latino | 48 | 58 | 106
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 43 | 49 | 92
  White | 3 | 13 | 16
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 54 | 64 | 118

OUTCOME MEASURES:

1. Primary Outcome: Cocaine Use as Assessed by Proportion of Visits (Excluding Excused Absences) With Cocaine-negative Urine Drug Screen
Description: Urine is assessed for levels of the cocaine metabolite benzoylecgonine (BE), and the drug screen is considered positive for cocaine use if BE level is ≥ 150 ng/mL.
Time Frame: 4 weeks
Population: Using a modified intention-to-treat plan, data are reported for all participants who completed at least one visit after randomization.
Measure: Mean (Standard Deviation); unit: proportion of visits
Units Other Than Participants: visits
Arm/Group | Phase 1: ACT Plus CM | Phase 1: DC Plus CM
Number analyzed (Participants) | 53 | 57
Number analyzed (visits) | 627 | 648
proportion of visits | 0.31 (0.36) | 0.24 (0.34)

2. Primary Outcome: Cocaine Use as Assessed by Proportion of Visits (Excluding Excused Absences) With Cocaine-negative Urine Drug Screen
Description: as for outcome 1
Time Frame: 12 Weeks
Population: Data are reported for all participants who started phase 2.
Measure: Mean (Standard Deviation); unit: proportion of visits
Units Other Than Participants: visits
Arm/Group | ACT Plus CM | ACT Plus CM, With Placebo | ACT Plus CM, With Modafinil | DC Plus CM | DC Plus CM, With Placebo | DC Plus CM, With Modafinil
Number analyzed (Participants) | 14 | 17 | 19 | 10 | 23 | 20
Number analyzed (visits) | 486 | 593 | 703 | 349 | 808 | 701
proportion of visits | 0.67 (0.24) | 0.22 (0.24) | 0.12 (0.12) | 0.70 (0.32) | 0.12 (0.15) | 0.10 (0.15)

3. Secondary Outcome: Cocaine Use as Indicated by Proportion of Days of no Cocaine Use as Assessed by Timeline Follow-back
Description: Timeline Followback (TLFB) is a method to assess of cocaine use that involves asking study participants to self-report their cocaine use over the past week.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: proportion of days
Arm/Group | Phase 1: ACT Plus CM | Phase 1: DC Plus CM
Number analyzed (Participants) | 53 | 57
proportion of days | 0.70 (0.23) | 0.66 (0.27)

4. Secondary Outcome: Cocaine Use as Assessed by Proportion of Days of no Cocaine Use as Assessed by Timeline Follow-back
Description: as for outcome 3
Time Frame: 12 Weeks
Population: Data are reported for all participants who started phase 2.
Measure: Mean (Standard Deviation); unit: proportion of days
Arm/Group | ACT Plus CM | ACT Plus CM, With Placebo | ACT Plus CM, With Modafinil | DC Plus CM | DC Plus CM, With Placebo | DC Plus CM, With Modafinil
Number analyzed (Participants) | 14 | 17 | 19 | 10 | 23 | 20
proportion of days | 0.83 (0.10) | 0.58 (0.31) | 0.70 (0.16) | 0.88 (0.11) | 0.63 (0.27) | 0.64 (0.27)

ADVERSE EVENTS:
Time Frame: 12 weeks
Groups:
- Phase 1: Acceptance and Commitment Therapy (ACT) Plus Contingency Management (CM) Only: In phase 1 (weeks 1-4), ACT plus CM for cocaine use will be administered to help decrease experiential avoidance while increasing acceptance and willingness to experience unpleasant thoughts, feelings, and physical symptoms.
- Phase 1: Drug Counseling (DC) Plus Contingency Management (CM) Only: In phase 1 (weeks 1-4), DC plus CM for cocaine use will be administered to help educate patients about important concepts in addiction recovery.
- Phase 2: ACT Plus CM Only: In phase 2 (weeks 5-12), ACT plus CM for cocaine use will continue to be administered.
- Phase 2: ACT Plus CM, With Placebo: In phase 2 (weeks 5-12), ACT plus CM for cocaine use will continue to be administered and participants will also receive placebo.
- Phase 2: ACT Plus CM, With Modafinil: In phase 2 (weeks 5-12), ACT plus CM for cocaine use will continue to be administered and participants will also receive modafinil.
- Phase 2: DC Plus CM Only: In phase 2 (weeks 5-12), DC plus CM for cocaine use will continue to be administered.
- Phase 2: DC Plus CM, With Placebo: In phase 2 (weeks 5-12), DC plus CM for cocaine use will continue to be administered and participants will also receive placebo.
- Phase 2: DC Plus CM, With Modafinil: In phase 2 (weeks 5-12), DC plus CM for cocaine use will continue to be administered and participants will also receive modafinil.
Arm/Group | Phase 1: Acceptance and Commitment Therapy (ACT) Plus Contingency Management (CM) Only | Phase 1: Drug Counseling (DC) Plus Contingency Management (CM) Only | Phase 2: ACT Plus CM Only | Phase 2: ACT Plus CM, With Placebo | Phase 2: ACT Plus CM, With Modafinil | Phase 2: DC Plus CM Only | Phase 2: DC Plus CM, With Placebo | Phase 2: DC Plus CM, With Modafinil
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/64 | 0/14 | 0/17 | 0/19 | 0/10 | 0/23 | 0/20
Serious Adverse Events (participants affected / at risk) | 3/54 | 1/64 | 0/14 | 0/17 | 0/19 | 1/10 | 0/23 | 3/20
Other Adverse Events (participants affected / at risk) | 11/54 | 14/64 | 2/14 | 10/17 | 8/19 | 0/10 | 10/23 | 14/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: Acceptance and Commitment Therapy (ACT) Plus Contingency Management (CM) Only (N=54) | Phase 1: Drug Counseling (DC) Plus Contingency Management (CM) Only (N=64) | Phase 2: ACT Plus CM Only (N=14) | Phase 2: ACT Plus CM, With Placebo (N=17) | Phase 2: ACT Plus CM, With Modafinil (N=19) | Phase 2: DC Plus CM Only (N=10) | Phase 2: DC Plus CM, With Placebo (N=23) | Phase 2: DC Plus CM, With Modafinil (N=20)
Domestic Violence/Abuse (Social circumstances) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomach Flu (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal Ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthma Attack (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Symptoms of Congestive Heart Failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: Acceptance and Commitment Therapy (ACT) Plus Contingency Management (CM) Only (N=54) | Phase 1: Drug Counseling (DC) Plus Contingency Management (CM) Only (N=64) | Phase 2: ACT Plus CM Only (N=14) | Phase 2: ACT Plus CM, With Placebo (N=17) | Phase 2: ACT Plus CM, With Modafinil (N=19) | Phase 2: DC Plus CM Only (N=10) | Phase 2: DC Plus CM, With Placebo (N=23) | Phase 2: DC Plus CM, With Modafinil (N=20)
Drowsiness (General disorders) | 0 (0) | 1 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (5)
Not Sleeping Well (General disorders) | 1 (1) | 2 (3) | 1 (1) | 2 (4) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Headache (General disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nervousness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blurry Vision (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Tremor (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomach Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle Aches (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (6)
Heart Racing (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (10) | 0 (0)
Increased Urination (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (12) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Change in Sexual Function (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weakness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Sweating (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dry Mouth (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 2 (9)
Difficulty Walking (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Skin Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (7)
Swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Loss of Appetite (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-15): https://cdn.clinicaltrials.gov/large-docs/12/NCT02896712/Prot_SAP_000.pdf